CLINICAL TRIAL: NCT04575649
Title: Neurodevelopmental Outcomes and Growth in Infants With Congenital Gastrointestinal Anomalies Requiring Neonatal Surgery
Acronym: NOGINS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1910-132
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Gastrointestinal Disease
Keywords: Body composition
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gastrointestinal anomalies — Infants born late preterm (at or above 35 weeks gestation) and term infants admitted to the NICU with congenital gastrointestinal anomalies, including gastroschisis, omphalocele, esophageal and bowel artesias, tracheoesophageal fistulas, Hirschsprung's disease, or congenital diaphragmatic hernias.

SUMMARY:
Infants with congenital gastrointestinal anomalies (CGIA) experience multiple physiologic stressors, including neonatal surgery, early in life during an essential time of growth and development. Early physiologic stressors such as inadequate nutrition have been linked to altered growth patterns and neurodevelopmental delays later in life. In other groups of at-risk infants, early body composition measurements can be used as predictors of long-term health outcomes more so than weight and length alone. The primary objective of this study is to determine if body composition changes in early life are predictive of neurodevelopmental outcomes among infants with CGIA. The secondary objective is to determine if infants with CGIA have altered body composition over time when compared with healthy infants. The investigators propose a prospective, observational study of infants with CGIA, including detailed chart review, body composition measurements, and neurodevelopmental testing at follow-up. If a correlation between body composition measurements and neurodevelopmental outcomes is established in this population, the addition of body composition measurement to standard of care in the neonatal intensive care unit and in follow-up care could allow for further optimization of overall health and development of this vulnerable pediatric population through earlier detection of growth alterations and informed interventions.

DETAILED DESCRIPTION:
Infants with congenital gastrointestinal anomalies (CGIA) including gastroschisis, omphalocele, esophageal and bowel atresias, tracheoesophageal fistulas, Hirschsprung's disease, and congenital diaphragmatic hernias, account for ~7 in 10,000 live births. Early in life, these infants undergo major surgery under general anesthesia followed by a prolonged period of inadequate nutrition, exposure to post-operative pain medications and antibiotics, and parental separation. Despite exposure to these risk factors for future growth failure and neurodevelopmental delay, growth and neurodevelopmental outcomes have not been well described in this group of at-risk infants. Preliminary findings in preschool-age children with CGIA suggest that these children have slower speed of processing compared to healthy children and that increased fat-free mass (FFM) at preschool age is associated with higher cognitive test scores. However, no studies to date have described the longitudinal relationship between growth, body composition, nutrition, inflammation, and neurodevelopmental outcomes in infants with CGIA. To address this research gap, the investigators propose to conduct a prospective cohort study enrolling infants with CGIA to measure their growth and development over time. Infant growth and body composition will be measured at or near term and at 4 months corrected age.

The investigators hypothesize that infants with CGIA will undergo a period of rapid catch-up growth early in life, and infants who demonstrate better catch-up growth will have better neurodevelopmental outcomes compared to infants that do not experience catch-up growth. At 4 months corrected age, early neurologic outcomes will be measured using event related potentials (ERP). Clinical information including nutrient intake, inflammatory markers, and medications received will be gathered throughout the neonatal intensive care unit (NICU) hospitalization to assess the impact physiologic stressors have on changes in body composition and cognitive outcomes.

The objective of this study is to determine the impact of early nutrition, inflammation, physiologic stress, growth, and body composition on later neurodevelopmental outcomes in infants requiring neonatal surgery for CGIA.

Specific aims include:

Aim 1. To determine if infants with CGIA requiring neonatal surgery have altered body composition growth patterns compared to healthy infants.

Aim 1a. To determine if early physiologic stress and/or malnutrition are associated with altered body composition in infants with CGIA compared to healthy infants.

Hypothesis: CGIA infants with increased early nutritional intake and decreased inflammation will have greater FFM gains and more appropriately mimic the growth of healthy comparison infants.

Aim 2. To determine if FFM gains in infancy are associated with improved neurodevelopmental outcomes among infants with CGIA.

Hypothesis: Greater FFM gains from birth to 4 months corrected age will be associated with faster speed of processing and better recognition memory among infants with CGIA.

The investigators hypothesize that early exposure to physiologic stressors impact the framework of the developing brain leading to long-lasting changes in development and that FFM accretion is an important biomarker of long-term outcomes for this population. The investigators hope to discover methods to better identify those infants at risk for poor neurodevelopmental outcomes and provide improved recommendations regarding nutritional and educational interventions that will ensure these infants achieve their full potential. These findings could also be used to encourage local and national NICU follow-up programs to expand beyond the follow-up of preterm infants to include high-risk populations such as infants born with CGIA. In addition, this proposed study could greatly impact community population health by optimizing growth and neurodevelopmental outcomes in children previously hospitalized in NICUs.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm (at or above 35 weeks gestation) and term infants
* Admitted to the NICU
* Diagnosed with congenital gastrointestinal anomalies, defined as gastroschisis, omphalocele, esophageal and bowel atresias, tracheoesophageal fistulas, Hirschsprung's disease, or congenital diaphragmatic hernias.

Exclusion Criteria:

* Infants born before 35 weeks gestation
* Infants with cardiac defects requiring intervention
* Infants with known chromosomal abnormalities that affect growth or cognition
* Infant born to families that are non-English speaking due to lack of interpreter services available

Ages: 0 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted to the NICU at University of Minnesota Masonic Children's Hospital, Children's Minnesota - St. Paul, or Children's Minnesota - Minneapolis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth | At term equivalence and at 4 months corrected age
  Anthropometric and body composition measurements

SECONDARY OUTCOMES:
Neurodevelopment | At 4 months
  Neurodevelopmental measures, defined as speed of processing, as associated with body composition

CONTACTS AND LOCATIONS:
Overall Officials: Erin Plummer, MD, Principal Investigator — Children's Minnesota
Locations (1):
- Children's Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided